CLINICAL TRIAL: NCT03845101
Title: SoREAL- a Randomized Clinical Trial
Brief Title: CBT Versus CBT With Virtual Reality Exposure for Social Anxiety Disorder and Agoraphobia
Acronym: SoREAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NNF17OC0027780
Record Dates: First submitted 2019-01-21; First posted 2019-02-19 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Social Anxiety Disorder; Agoraphobia
Keywords: Social anxiety; Virtual Reality; Virtual Reality Exposure Therapy; RCT; Social Phobia; Agoraphobia
MeSH Terms: conditions — Phobia, Social; Agoraphobia | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT in virtuo (Experimental): Receives CBT in group format with Virtual Reality Exposure Therapy
  Interventions: Behavioral: CBT with virtual reality exposure therapy
- CBT in vivo (Active Comparator): Active comparator, receives CBT in group format. Treatment as usual.
  Interventions: Behavioral: CBT in vivo

INTERVENTIONS:
Behavioral: CBT with virtual reality exposure therapy — The patients receiving the in virtuo exposure will be immersed using an Oculus Go head-mounted display, enabling viewing of 360° spherically camera recorded VR environments. The VR scenarios will thus be high-resolution 360° stereoscopic films, that are played around the viewer. For ease of use, the individual videos will be administered from an app that has been designed to be as intuitive to operate as possible. The patient will only have to put on the headset, adjust the focus and choose the desired environment by looking at it in the app. 360° video was chosen because it gives the most photorealistic visuals, while also being the cheapest to produce. The downside is that it does not allow direct user-interaction (e.g. the viewer cannot affect the environment in any way). To circumvent this, there are multiple junctions throughout the films where the actors will talk directly and unsolicited to the viewer while also allowing time for the viewer to respond.
  Arms: CBT in virtuo
Behavioral: CBT in vivo — The therapeutic intervention is manual-based cognitive-behavioral CBT group therapy adapted from the approach of Turk, Heimberg & Magee and Graske & Barlow with worksheets from Arendt & Rosenberg and inspiration from Bouchard et al. The treatment will consist of 14 weekly two-hour group sessions following the manual to ensure equal and uniform treatment for every patient throughout the study. Concurrent psychopharmacological treatment is allowed in both intervention arms.
  Arms: CBT in vivo

SUMMARY:
Introduction: Anxiety disorders have a high lifetime prevalence, early-onset, and long duration or chronicity. Exposure therapy is considered one of the most effective elements in cognitive behavioral therapy (CBT) for anxiety, but in vivo exposure can be challenging to access and control, and is sometimes rejected by patients because they consider it too aversive. Virtual reality allows flexible and controlled exposure to challenging situations in an immersive and protected environment.

Aim: The SoREAL-trial aims to investigate the effect of group cognitive-behavioral therapy (CBT-in vivo) versus group cognitive behavioral therapy with virtual reality exposure (CBT-in virtuo) for patients diagnosed with social anxiety disorder and/or agoraphobia, in mixed groups.

Methods & Analysis: The design is an investigator-initiated randomized, assessor-blinded, parallel-group and superiority-designed clinical trial. Three hundred two patients diagnosed with social anxiety disorder and/or agoraphobia will be included from the regional mental health centers of Copenhagen and North Sealand and the Northern Region of Denmark. All patients will be offered a manual-based 14-week cognitive behavioral group treatment program, including eight sessions with exposure therapy. Therapy groups will be centrally randomized with concealed allocation sequence to either CBT-in virtuo or CBT-in vivo. Patients will be assessed at baseline, post-treatment and one-year follow-up by treatment blinded researchers and research assistants. The primary outcome will be diagnosis-specific symptoms measured with the Liebowitz Social Anxiety Scale for patients with social anxiety disorder and the Mobility Inventory for Agoraphobia for patients with agoraphobia. Secondary outcome measures will include depression symptoms, social functioning, and patient satisfaction. Exploratory outcomes will be substance and alcohol use, working alliance and quality of life.

Ethics and dissemination: The trial has been approved by the research ethics committee in the Capital Region of Denmark. All results, positive, negative as well as inconclusive, will be published as quickly as possible and still in concordance with Danish law on the protection of confidentially and personal information. Results will be presented at national and international scientific conferences.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling diagnostic criteria for social anxiety disorder (ICD-code: F40.1) and/or Agoraphobia (ICD-code: 40.0)
* Age 18-75 years
* Sufficient knowledge of the Danish language
* Informed consent

Exclusion Criteria:

* Alcohol or drug dependence (ICD-code: F10-19.20-26).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2024-04-09 (Estimated); Study Completion 2024-04-09 (Estimated)

PRIMARY OUTCOMES:
Change in symptom severity of primary diagnosis | Between 30 to 1 day(s) before treatment, between 0 and 14 days after treatment ends and between 365 to 395 days after first assesment.
  Total scores on the Liebowitz Social Anxiety Scale (LSAS) for patients with social anxiety disorder and the Mobility Inventory for Agoraphobia (MIA) for patients with Agoraphobia measured pre-treatment, post-treatment and at one-year follow-up converted to the 'Percentage of Maximum Possible Score' (POMP) and averaged within treatment arms. POMP calculations can bring differently measured items to the same metric and do not change the multivariate distribution and covariance matrix of the transformed variables.
  Ranges from 0 to 100. Higher is worse.

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale, 6 item score | Between 30 to 1 day(s) before treatment, between 0 and 14 days after treatment ends and between 365 to 395 days after first assesment.
  Measures symptoms of depression for the last 3 days.Total score will be measured. Ranges from 0 to 22. Higher is worse.
Change in Brief Version of the Fear of Negative Evaluation Scale score | Between 30 to 1 day(s) before treatment, between 0 and 14 days after treatment ends and between 365 to 395 days after first assesment.
  Self-report, total score is measured, ranging from 12 to 60. Higher is worse.
Change in Work and Social Adjustment Scale score | Between 30 to 1 day(s) before treatment, between 0 and 14 days after treatment ends and between 365 to 395 days after first assesment.
  Self-report. Total score is measured, ranging from 0 to 40. Higher is better.
Client Satisfaction Questionnaire | Measured between 0 and 14 days after treatment ends
  Measures satisfaction with treatment. Total score is measured, ranging from 8 to 32. Higher is better. Self-report.
Change in WHO Well-Being Index 5 items, score | Between 30 to 1 day(s) before treatment, between 0 and 14 day(s) after treatment ends and between 365 to 395 days after first assesment.
  Measures overall quality of life. Total score is measured. Ranges from 0 to 25. Higher is better. Self-report.
Treatment response on social anxiety disorder symptoms | Between 0 and 14 day(s) after treatment ends and between 365 to 395 days after first assesment.
  Liebowitz Social Anxiety Scale total score below 50 or a 15 points drop.
  Ranges from 0 to 144. Higher is worse.
Treatment response on agoraphobia symptoms | Between 0 and 14 day(s) after treatment ends and between 365 to 395 days after first assesment.
  Mobility Inventory for Agoraphobia total score below 2 or a 0.5 points drop
  Ranges from 0 to 5. Higher is worse.
Remission from social anxiety disorder | Between 0 and 14 day(s) after treatment ends and between 365 to 395 days after first assesment.
  Liebowitz Social Anxiety Scale total score below 25 and not qualifying for social anxiety disorder as measured using the MINI-7.
  Ranges from 0 to 144. Higher is worse.
Remission from agoraphobia | Between 0 and 14 day(s) after treatment ends and between 365 to 395 days after first assesment.
  MIA total score below 1.5 and not qualifying for agoraphobia as measured using the MINI-7.
  Ranges from 0 to 5. Higher is worse.

OTHER OUTCOMES:
Change in Personal and Social Performance Scale score | Between 30 to 1 day(s) before treatment, between 0 and 14 day(s) after treatment ends and between 365 to 395 days after first assesment.
  Measured as total score. Ranges from 0 to 100. Higher is better. Self-report.
Change in Alchohol and drug (legal and illegal) use | Between 30 to 1 day(s) before treatment, between 0 and 14 day(s) after treatment ends and between 365 to 395 days after first assesment.
  Measured using the Time Line Follow Back interview, in which you systematically go through every day for the last 4 weeks recording any alcohol and drug (legal and illegal) consumption. Will be scored in units of 12 grams of alcohol and in grams of substance consumed. Less consumed alchohol and substance will be considered better.
Change in General Self Efficacy Scale Score | Between 30 to 1 day(s) before treatment, between 0 and 14 day(s) after treatment ends and between 365 to 395 days after first assesment.
  Measures general belief in ones own capabilities. Self-report. Total score is measured. Ranges from 10 to 40. Higher is better.
Working Alliance Inventory | Measured between 0 and 14 days after treatment ends.
  Measured the experience of alliance between the client and the therapist(s). Self-report. Total score is measured. Ranges from 12 to 60. Higher score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Merete Nordentoft, Principal Investigator — Mental Health Centre Copenhagen (CORE)
Locations (5):
- Denmark (5):
  - Psykoterapeutisk Klinik, Nannasgade, Copenhagen, Captial Region of Denmark
  - Psykoterapeutisk Ambulatorium, Brøndby, Copenhagen
  - Psykoterapeutisk klinik, Frederiksberg, Frederiksberg, Copenhagen
  - Psykoterapeutisk Center Stolpegård, Gentofte Municipality, Copenhagen
  - Ambulatorium for Angst og Tvangssygdomme, Aalborg

IPD SHARING:
Plan to Share IPD: Yes
After completed analyses and publication, all depersonalised individual patient data will be transferred to The Danish National Archives and made available for other researchers upon reasonable request and with permission of The Danish National Archives.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The current policy of The Danish National Archives is to keep data stored securely indefinitely.
  Data will be transfered The Danish National Archives after completed analyses and publication. However, this can take a maximum of 10 years, after which data must be refered to the National Archives.
Access Criteria: Reasonable request and permission of The Danish National Archives.

REFERENCES:
- [Background] Turk CL, Heimberg RG, Magee L. Social anxiety disorder. In: Barlow DH, editor. Clin Handb Psychol Disord A step-by-step Treat Man. London: Guilford Press; 2008. p. 123-63.
- [Background] Graske MG, Barlow DH. Panic Disorder and Agoraphobia. In: Barlow DH, editor. Clin Handb Psychol Disord. 4th ed. New York: The Guilford Press; 2008. p. 1-65.
- [Background] Rosenberg NK, Mørck MM, Arendt M. Kognitiv terapi. Nyeste udvikling. Kogn Ter Nyeste Udvikl. 2012.
- [Background] Bouchard S, Robillard G, Larouche S, Loranger C. Description of a treatment manual for in virtuo exposure with specific phobia. Virtual Real Psychol Med Pedagog Appl. 2012;81-108.
- [Derived] Arnfred B, Bang P, Hjorthoj C, Christensen CW, Stengaard Moeller K, Hvenegaard M, Agerskov L, Krog Gausboel U, Soe D, Wiborg P, Smith CIS, Rosenberg N, Nordentoft M. Group cognitive behavioural therapy with virtual reality exposure versus group cognitive behavioural therapy with in vivo exposure for social anxiety disorder and agoraphobia: a protocol for a randomised clinical trial. BMJ Open. 2022 Feb 2;12(2):e051147. doi: 10.1136/bmjopen-2021-051147. PMID 35110313